CLINICAL TRIAL: NCT00881023
Title: A Multicenter, Randomized, Pivotal Study to Evaluate the Safety and Efficacy of the Cartilage Autograft Implantation System (CAIS) for the Surgical Treatment of Articular Cartilage Lesions of the Knee
Brief Title: Cartilage Autograft Implantation System (CAIS) for the Repair of Knee Cartilage Through Cartilage Regeneration
Acronym: CAIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated because of very low enrollment rate.
Sponsor: DePuy Mitek (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-CAIS-05; IDE # 11803 (Other: FDA); NCT00595803 (obsolete NCT alias); NCT01508442 (obsolete NCT alias)
Record Dates: First submitted 2009-04-10; First posted 2009-04-14 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Defect of Articular Cartilage; Osteochondritis Dissecans
MeSH Terms: conditions — Osteochondritis Dissecans | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Randomized to Microfracture
  Interventions: Procedure: Microfracture
- 2 (Experimental): Randomized to Device
  Interventions: Device: Cartilage Autograft Implantation System
- 3 (Experimental): Non-randomized with lesion greater than 6cmˆ2
  Interventions: Device: Cartilage Autograft Implantation System

INTERVENTIONS:
Procedure: Microfracture — The microfracture procedure is a standard method for treatment of cartilage damage in which the surgeon will clean the site of your cartilage damage and then will make several small holes in your bone to stimulate your bone marrow with the intention to repair the damaged area with new cartilage tissue
  Arms: 1
Device: Cartilage Autograft Implantation System — A surgical treatment of damaged knee cartilage using the subject's own healthy cartilage obtained from a non-weight or low weight-bearing region
  Arms: 2; 3

SUMMARY:
The Cartilage Autograft Implantation System (CAIS) is designed as a single surgical treatment of damaged knee cartilage using the subject's own healthy cartilage obtained from a non-weight or low weight-bearing region. CAIS is indicated for the repair of articular cartilage lesions and osteochondritis dissecans (OCD) of the knee through cartilage regeneration.

DETAILED DESCRIPTION:
The Cartilage Autograft Implantation System (CAIS) is a kit of devices that utilizes morselized autologous hyaline cartilage harvested arthroscopically, affixed onto a synthetic, resorbable implant using a fibrin sealant and implanted in a single surgical procedure. The system is designed as a surgical treatment of damaged knee cartilage using the subject's own healthy cartilage obtained from a non-weight or low weight-bearing region.

ELIGIBILITY:
Inclusion Criteria:

* A male or female 18 to 55 years of age,
* Has 1 or 2 focal chondral lesions, that require repair, per index knee presenting with moderate to severe knee pain. Each lesion is ≤6 mm in depth and has an area of ≥1 cm2 and ≤10 cm2. Arthroscopic confirmation indicates that the lesions are either a non-OCD lesion between grades I and III (D) or an OCD lesion between grades I and IV(A)
* Prior failed chondral treatment is allowed if the procedure occurred > 6 months for debridement and lavage or > 1 year for marrow stimulation techniques.

Exclusion Criteria:

* Have more than 2 chondral lesions on the index knee,
* Bipolar lesions on the index knee,
* Greater than 5 degrees of malalignment,
* Require bilateral surgery
* Have a diagnosis of clinical and/or radiographic disease of the index joint.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2010-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To determine the safety and efficacy of CAIS compared to microfracture at 24 months post-treatment, with the primary efficacy assessment based on an analysis of superiority of CAIS to microfracture for reduction in knee pain and improvement in function | 24 Months

SECONDARY OUTCOMES:
To determine the safety of CAIS through 48 months | 48 Months

CONTACTS AND LOCATIONS:
Overall Officials: Brooks Story, PhD, Study Director — DePuy Synthes Mitek Sports Medicine
Locations (29):
- United States (27):
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - MWMC Bentonville Hospital, Bentonville, Arkansas
  - CORE Orthopaedic Medical Center, Encinitas, California
  - Santa Monica Orthopaedic Group, Santa Monica, California
  - Southern California Orthopaedic Group, Van Nuys, California
  - JDP Medical Research, LLC, Denver, Colorado
  - Shrock Orthopedic Research, Fort Lauderdale, Florida
  - Andrews Institute, Gulf Breeze, Florida
  - Florida Orthopaedics Institute and Research Foundation, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - OrthoIndy, Indianapolis, Indiana
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Harvard Vanguard / New England Baptist Hospital, Chestnut Hill, Massachusetts
  - UMass Medical Center - Orthopedic Research, Worcester, Massachusetts
  - TRIA Orthopaedic Center, Bloomington, Minnesota
  - University of Missouri, Columbia, Missouri
  - Rothman Institute, Egg Harbor, New Jersey
  - University Orthopaedic Group LLC, New Brunswick, New Jersey
  - New York University School of Medicine, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Orlin & Cohen Orthopedic Group, Rockville Centre, New York
  - Ohio State University, Columbus, Ohio
  - Orthopaedic Research Foundation of the Carolinas, Greenville, South Carolina
  - OrthoMemphis, PC, Memphis, Tennessee
  - Basin Orthopedic Surgical Specialists, Odessa, Texas
  - Richmond Bone & Joint Clinic, P.A., Sugar Land, Texas
  - University of Virginia, Charlottesville, Virginia
- Canada (2):
  - Royal Columbian Hospital, New West Minster, British Columbia
  - Fowler Kennedy Sports Medicine Clinic, New West Minister, Ontario

IPD SHARING:
Plan to Share IPD: No
These data will not be used in support of an FDA submission, and the product will not be commercialized. As such, there is no plan to share the IPD.